CLINICAL TRIAL: NCT07016958
Title: Effects of Carbohydrate Counting Training Versus Standard Nutritional and Medical Therapy on Glycemic Control and Sarcopenia in Type 2 Diabetes: A Randomized Controlled Trial
Brief Title: Carbohydrate Counting Training in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Funda GARGACI TUNCER, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IMU- SBE-FGT-01
Record Dates: First submitted 2025-05-31; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus Type 2; Sarcopenia
Keywords: Diabetes; carbohydrate; glycemic control; insulin; sarcopenia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sarcopenia; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: There are two groups: training and control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): The training group received advanced carbohydrate counting training in addition to standard medical and medical nutrition therapy.
  Interventions: Behavioral: Carbohydrate Counting Training
- Control Group (No Intervention): The control group continued standard medical and medical nutrition therapy only.

INTERVENTIONS:
Behavioral: Carbohydrate Counting Training — Advanced Carbohydrate Counting Training is a meal planning training where individuals can calculate the amount of carbohydrates in foods based on their portion sizes, and the insulin doses they need to take based on their plasma glucose levels and the amount of carbohydrates they consume.
  Arms: Training Group

SUMMARY:
This study aimed to evaluate the efficacy of carbohydrate counting in individuals with type 2 diabetes receiving intensive insulin therapy. In addition, the sarcopenia status in this patient group and the effect of carbohydrate counting on sarcopenia were also evaluated.

DETAILED DESCRIPTION:
Participants with type 2 diabetes receiving intensive insulin treatment were randomized and divided into 2 groups: education and control groups. Participants in the control group continued their standard medical and medical nutrition treatments. Participants in the training group received advanced carbohydrate counting training consisting of 3 sessions in addition to standard medical and medical nutrition therapy. The measurements of the participants in the training and control groups were repeated three times at the beginning of the study, in the 12th week and in the 24th week of the study.

A questionnaire form containing sociodemographic information was completed by face-to-face interview method. In addition, biochemical (HbA1c, fasting plasma glucose (FPG), C peptide, total cholesterol, HDL, LDL, triglyceride, estimated glomerular filtration rate) and anthropometric and body composition (weight-height, BMI, fat mass, fat ratio, muscle mass, lean tissue mass, waist circumference), hand grip strength and blood pressure measurements of the patients were taken at the beginning, 12th week and 24th week of the study.

In addition, a 24-hour retrospective food consumption record was applied to evaluate the energy and nutrient intakes. The calculation of the energy, macro and micro-nutrient intakes of the participants was carried out using the Turkish Nutrition Database Ebispro for Windows program (version 7.2)

ELIGIBILITY:
Inclusion Criteria:

* A history of type 2 diabetes mellitus
* Using insulin for more than one year
* Being over 18 years old
* Receiving basal and bolus insulin treatment
* Not having received carbohydrate counting training before
* Not receiving treatment with sulfanylurea drugs from oral anti-diabetics.

Exclusion Criteria:

* Being pregnant or breastfeeding or planning a pregnancy during the study period,
* Discontinuing insulin treatment during the study period
* Having active proliferative retinopathy, severe nephropathy, severe or newly diagnosed cardiac disease within 6 months or stage III-IV heart failure,
* Having dementia or psychosis and cognitive impairment,
* Receiving glucocorticoid treatment, being fed enterally or parenterally and receiving nutrition treatment due to another/concomitant disease, having end-stage renal or hepatic/ renal disease (other than proteinuria)
* Having liver disease/microangiopathy diseases
* Having clinical cancer, chronic respiratory disease or amputations,
* Having any disease or condition that would prevent completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
HbA1c (%) | Baseline, week 12 and week 24
  HbA1c levels of the participants were performed in the Biochemistry Laboratory of Fatih Sultan Mehmet Training and Research Hospital. The individuals participating in the study were asked to give blood in the morning after 10-12 hours of fasting after dinner. HbA1c levels were measured by high-performance liquid chromatography (HPLC) method. The statistical analysis of the data obtained from the study was evaluated using the IBM SPSS Statistics (version 22.0) package program.
Plasma Glucose Levels | Baseline, week 12 and week 24
  Plasma glucose levels of the participants were performed in the Biochemistry Laboratory of Fatih Sultan Mehmet Training and Research Hospital. The individuals participating in the study were asked to give blood in the morning after 10-12 hours of fasting after dinner. Plasma glucose levels were analyzed by hexokinase method in colorimetric-spectrophotometric Aeroset (Roche Hitachi cobas 6000) autoanalyzer. The statistical analysis of the data obtained from the study was evaluated using the IBM SPSS Statistics (version 22.0) package program.
Muscle Strength | Baseline, week 12, week 24
  It was used for the evaluation of sarcopenia. The participants' hand grip strength was measured three times with a digital hand dynamometer (CAMRY-EH101, USA) and the mean value in kg was calculated. The statistical analysis of the data obtained from the study was evaluated using the IBM SPSS Statistics (version 22.0) package program.
Skeletal muscle mass | Baseline, week 12, week 24
  It was used for the evaluation of sarcopenia. Skeletal muscle mass data obtained from the BIA measurement results and skeletal muscle according to the height obtained from this data were calculated by dividing the skeletal muscle mass by the square of the height.The statistical analysis of the data obtained from the study was evaluated using the IBM SPSS Statistics (version 22.0) package program.
Physical performance | Baseline, week 12 and week 24
  It was used for the evaluation of sarcopenia. In the timed walk-up test, the patient is asked to get up from the chair, walk at a normal walking speed on a flat surface of 3 meters, turn around, walk back and sit back in the chair. The time between the patient getting up from the chair, walking and sitting down again is recorded and the patient's dynamic balance during walking is also evaluated. The statistical analysis of the data obtained from the study was evaluated using the IBM SPSS Statistics (version 22.0) package program.

SECONDARY OUTCOMES:
Blood lipid levels | Baseline, week 12 and week 24
  Blood lipid levels of the participants were performed in the Biochemistry Laboratory of Fatih Sultan Mehmet Training and Research Hospital. The individuals participating in the study were asked to give blood in the morning after 10-12 hours of fasting after dinner. total cholesterol, HDL and triglyceride levels were analyzed by enzymatic colorimetric method. LDL levels were calculated using the Fridewald equation. The statistical analysis of the data obtained from the study was evaluated using the IBM SPSS Statistics (version 22.0) package program.
Hypoglicemia Period | Baseline, week 12 and week 24
  It refers to the periods of hypoglycemia that individuals experience within a month. This data was asked of patients when their measurements were taken. The statistical analysis of the data obtained from the study was evaluated using the IBM SPSS Statistics (version 22.0) package program.
Total Insulin Dose | Baseline, week 12 and week 24
  It is the insulin dose that individuals need to take to keep their plasma glucose levels at ideal levels during the day. This data was asked of the patients while their measurements were being taken and was verified from the patient record system in the hospital.The statistical analysis of the data obtained from the study was evaluated using the IBM SPSS Statistics (version 22.0) package program.
Daily Prandial Insulin | Baseline, week 12 and week 24
  It is the insulin dose that individuals should take before meals to keep their plasma glucose levels at an ideal level during the day. This data was asked of the patients while their measurements were being taken and was verified from the patient record system in the hospital. The statistical analysis of the data obtained from the study was evaluated using the IBM SPSS Statistics (version 22.0) package program.
Daily Basal Insulin | Baseline, week 12 and week 24
  It is the insulin dose that individuals need to take to keep their plasma glucose levels at ideal levels during the day. This data was asked of the patients while their measurements were being taken and was verified from the patient record system in the hospital. The statistical analysis of the data obtained from the study was evaluated using the IBM SPSS Statistics (version 22.0) package program.
Serum C peptide Levels | Baseline
  Serum C peptide levels were examined because insulin doses and carbohydrate counting were thought to affect training outcomes.Serum C peptide levels of the participants were performed in the Biochemistry Laboratory of Fatih Sultan Mehmet Training and Research Hospital. The individuals participating in the study were asked to give blood in the morning after 10-12 hours of fasting after dinner. Serum C peptide levels were determined by Enzyme-Linked Immunosorbent Assay (ELISA) method (Roche Hitachi cobas 6000) using a commercial kit in an autoanalyzer. The statistical analysis of the data obtained from the study was evaluated using the IBM SPSS Statistics (version 22.0) package program.
Glomerular filtration rate | Baseline, week 12, week 24
  Glomerular filtration rate of the participants were performed in the Biochemistry Laboratory of Fatih Sultan Mehmet Training and Research Hospital. The individuals participating in the study were asked to give blood in the morning after 10-12 hours of fasting after dinner. The statistical analysis of the data obtained from the study was evaluated using the IBM SPSS Statistics (version 22.0) package program.
Diastolic and Sistolic Blood Pressure | Baseline, week 12, week 24
  Blood pressure of the participants was measured with an automatic sphygmomanometer (SCIAN LD-533, Germany). Three repeated measurements were made on the right arm in the sitting position with the arm at the level of the heart and after a rest period of at least 10 minutes and the mean was calculated. The statistical analysis of the data obtained from the study was evaluated using the IBM SPSS Statistics (version 22.0) package program.
Waist circumference | Baseline, week 12 and week 24
  Anthropometric measurements of the participants were taken by a dietician. In waist circumference measurement, the midpoint between the bottom of the rib bone and the iliac crest was determined and the circumference of this area was measured with a tape measure. The statistical analysis of the data obtained from the study was evaluated using the IBM SPSS Statistics (version 22.0) package program.
Hyperglycemia period | Baseline, week 12 and week 24
  It refers to the periods of hyperglycemia that individuals experience within a month. This data was asked of patients when their measurements were taken. The statistical analysis of the data obtained from the study was evaluated using the IBM SPSS Statistics (version 22.0) package program.
Food consumption (energy and nutrients intake) | Baseline, week 12 and week 24
  A 24-hour retrospective food consumption record was applied to evaluate the energy and nutrient intakes. The calculation of the energy, macro and micro-nutrient intakes of the participants was carried out using the Turkish Nutrition Database Ebispro for Windows program (version 7.2) The statistical analysis of the data obtained from the study was evaluated using the IBM SPSS Statistics (version 22.0) package program.
Physical Activity Levels | Baseline, week 12 and week 24
  The International Physical Activity Questionnaire Short Form (IPAQ-SF) was used to determine physical activity levels. The statistical analysis of the data obtained from the study was evaluated using the IBM SPSS Statistics (version 22.0) package program.
Height | Baseline, week 12 and week 24
  Anthropometric measurements of the participants were taken by a dietician. The height of the participants was measured with a wall-type stadiometer with barefoot heels touching each other, arms hanging to the side, feet 45o apart and head in the Frankfort plan. The statistical analysis of the data obtained from the study was evaluated using the IBM SPSS Statistics (version 22.0) package program.
Body weight and body composition (fat weight, muscle weight, lean weight) | Baseline, week 12 and week 24
  Anthropometric measurements of the participants were taken by a dietician. Body weight and body composition were measured with TANITA BC-418MA bioelectrical impedance analyzer. The statistical analysis of the data obtained from the study was evaluated using the IBM SPSS Statistics (version 22.0) package program.
Body Mass Index | Baseline, week 12 and week 24
  BMI values of the participants were calculated based on weight and height measurement data. The statistical analysis of the data obtained from the study was evaluated using the IBM SPSS Statistics (version 22.0) package program.

CONTACTS AND LOCATIONS:
Overall Officials: Indrani KALKAN, Assoc. Prof., Study Director — Medipol University
Locations (1):
- Uskudar Diabetes Polyclinic of the Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/58/NCT07016958/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/58/NCT07016958/SAP_001.pdf